CLINICAL TRIAL: NCT05657015
Title: Lepidium Sativum Extract Versus Simvastatin as an Adjunctive Local Delivery Agents to Non-Surgical Periodontal Therapy: A Randomized Controlled Clinical Trial With Biochemical Analysis
Brief Title: Lepidium Sativum Extract Versus Simvastatin as an Adjunctive Local Delivery Agents to Non-Surgical Periodontal Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Local drug delivery
Record Dates: First submitted 2022-11-08; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Periodontitis
Keywords: In situ gel; High Performance Thic Layer Chromatography; Local Drug Delivery
MeSH Terms: conditions — Periodontitis | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: This study was designed to be a Randomized, Controlled, Triple-blinded, Phase (IV) clinical trial; the eligible participants were randomly allocated to one of the two comparative parallel groups; test and control group using computer-generated random tables (www.randomizer.org).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The phytochemicals were prepared by the pharmacist and coded so that the patients, researcher, and outcomes assessor were blinded to the type of intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lepidium sativum (Experimental): 15 participants 15 participants with localized stage II or III, and grade A periodontitis received about 2ml of locally delivered Lepidium sativum in situ gel with scaling and root surface debridement once at the beginning of the study
  Interventions: Drug: Lepidium Sativum
- simvastatin (Active Comparator): 15 participants with localized stage II or III, and grade A periodontitis received about 1.2% of locally delivered Simvastatin in situ gel with scaling and root surface debridement once at the beginning of the study
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Lepidium Sativum — 2 ml of LS in situ gel at baseline
  Other Names: Garden cress
  Arms: Lepidium sativum
Drug: Simvastatin — 1.2% of SMV in situ gel at baseline
  Arms: simvastatin

SUMMARY:
The objectives of this clinical study were to:

1. Assess the influence of Lepidium sativum in situ gel versus simvastatin gel on the clinical parameters in periodontitis patients as the primary objective.
2. Detect the effect of locally delivered Lepidium sativum and simvastatin gels on the nuclear factor kappa B (NF-κB) level in gingival crevicular fluid as the secondary objective.

DETAILED DESCRIPTION:
Periodontitis is a multifactorial inflammatory disease that is triggered by the accumulation of oral biofilm on the tooth surface, leading to progressive destruction of the periodontal supporting tissues including loss of clinical attachment level, alveolar bone resorption, and formation of periodontal pockets due to apical migration of junctional epithelium. It is characterized by microbially-associated, host-mediated inflammation that leads to loss of periodontal apparatus. The formation of a bacterial biofilm begins with gingival inflammation; however, the initiation and progression of periodontitis are based on microbiome dysbiotic ecological changes in response to nutrients from gingival inflammatory and tissue breakdown products. So periodontitis is defined as a chronic immuno-inflammatory disorder affecting all the tooth-supporting structures. The conventional treatment of periodontitis involves scaling and root surface debridement (RSD) which is the supra and subgingival mechanical debridement of the periodontal pockets. RSD is done either by manual instruments or by ultrasonic devices. Although it may be effective alone, it has limitations such as in the case of deep periodontal pockets, inaccessible areas, and severe status of the disease. Therefore, this treatment should be supported by adjunctive antibacterial agents to remove the residual bacteria. Antibacterial agents have been used along with mechanical debridement in the management of periodontal infection. For about the past 30 years, locally delivered, anti-infective pharmacological agents have been introduced to achieve this goal. Since the disease is confined to the periodontium, local delivery of the drug in the pocket itself is the best option. The pocket acts as a natural reservoir and provides easy access for the insertion of a medicinal device. Drug release and distribution throughout the pocket are provided by gingival crevicular fluid (GCF), which acts as the leaching medium. Also, significant drug levels can be maintained in the GCF for a prolonged duration. Local delivery drugs can overcome most of the adverse side effects of systemic agents. All these factors make intra-pocket drug delivery an ideal choice. Statins such as simvastatin (SMV) have been considered as an adjunct to non-surgical periodontal therapy. Statins were initially imported as cholesterol-reducing drugs, which is performed by hindering the 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase. Statins also have additional properties including; anti-inflammatory, anti-oxidant, anti-bacterial, and other pleiotropic effects such as blocking the release of pro-inflammatory mediators and matrix metalloproteinases (MMPs). Therefore, statins have been shown to promote bone formation and have proven to be effective in periodontal therapy. Nowadays, there are many researchers using plants as adjunctive therapy to the non-surgical periodontal treatment of disease because of their efficacy, safety, and therapeutic prominence. Lepidium sativum (LS) is one of the herbal products that is used daily without any regard for its benefits. It is an annual, edible herb that belongs to the family of Brassicaceae. It originated in Ethiopia and is found in many countries such as Saudi Arabia, India, and Egypt, and later in Europe. It had other names such as garden cress, halon, Hab Al-Rashad, and Thuffa. It is composed of seeds, leaves, and roots. All of its parts were important for medicinal effects. It has a peppery flavor so it can be used for homemade foods (as salads, and sandwiches), especially the leaves. The seeds can be used in many therapeutic domains as an anti-hyperglycemia, anti-hyperlipidemia, anti-diarrhea, anti-rheumatic, hepatoprotective, antioxidant, anti-inflammatory, and anti-microbial and in gastrointestinal, skin, and respiratory diseases, and some bone fractures healing. LS seeds contain many several phenols, minerals, proteins, fatty acids, vitamins, and carbohydrates. Because of its polyphenols composition, it has anti-microbial activity against several bacteria such as (P. auregenosa, S. aureus, and E. coli). The plant's antioxidative effect decreases the generation of reactive oxygen species on human cells and thus decreases the destruction of the disease. Oxygen stress plays an important role in the occurrence of many human diseases due to an increase in reactive oxygen species (ROS) production. Because of the anti-oxidant activity of the LS and cytoprotective effects, the pre-treatment with this plant can lead to inhibition of ROS generation. Tumor necrosis factor α (TNF-α), interleukin 6 and 10 (IL-6, IL-10), and nitric oxide (NO) are the pro-inflammatory mediators that play an important role in disease damage. Nuclear factor kappa B (NF-kB) also plays a role in inflammation by inducing the transcription of TNF-α on bacterial lipopolysaccharides (LPS). LPS may alter the anti-oxidative activity and enhance the production of inflammatory mediators. Therefore, the administration of LS seed extract will decrease the effectiveness of the bacteria and improve general health.

Due to the lack of studies that used LS as a therapeutic agent in periodontitis, the current study was performed to evaluate this plant's efficacy in the management of periodontitis. Furthermore, due to the pleiotropic effects of Simvastatin and Lepidium sativum, the present study was carried on to assess the influence of LS gel versus simvastatin gel as an adjunct to non-surgical periodontal therapy. Moreover, the effects of SMV and LS on the level of NF-κB in GCF were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ages ranging from 25 to 50 years old.
* Localized periodontitis, probing depth ≥5 mm. Less than 30% of teeth are involved.
* Both genders.
* Patients must be able to return for the recall visits and agreed to sign the written consent after a full explanation of the study.
* Systemically free according to the American Society of Anesthesiologists (ASA I).

Exclusion Criteria:

* Smokers
* Pregnant and lactating women or oral contraceptive usage
* Prisoners or abused individuals
* Unwilling patients to perform oral hygiene measures of plaque control.
* Patients with a history of allergy against any components of the two materials.
* Previous Periodontal treatment or any use of antibiotic/anti-inflammatory drugs within the last 6 months before the initiation of the study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Assess clinically the plaque index (PI) in periodontitis patients | Change at baseline (after 1 week from the last debridement) and after 3 months follow-up period
  Percentage of tooth surfaces with bacterial deposits. Plaque index scores were recorded at six sites per tooth (mesiobuccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual).The plaque index visually records the score such as 0,1,2, and 3 using the standard probe.
Asses clinically the mean sulcus bleeding index (MSBI) in periodontitis patients | Change at baseline (after 1 week from the last debridement) and after 3 months follow-up period
  Percentage of tooth surfaces with bleeding point sites on probing. Bleeding index scores were recorded at six sites (mesiobuccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual). The scores were recorded as 0,1,2,3,4, and 5.
Assess clinically the probing depth (PD) in periodontitis patients | Change at baseline (after 1 week from the last debridement) and after 3 months follow-up period
  The distance between the margin of the gingiva and the base of the pocket was recorded at four points (mesio-facial, mid-facial, disto-facial, and mid-lingual) to the nearest millimeter using the University of Michigan O' probe with Williams' graduations in conjunction with an occlusal stent for the standardization of readings. The probe was inserted parallel to the long axis of the tooth.
Assess clinically the clinical attachment level (CAL) in periodontitis patients | Change at baseline (after 1 week from the last debridement) and after 3 months follow-up period
  The CAL was measured in millimeters from the cemento-enamel junction (CEJ) to the base of the pocket using the University of Michigan O' probe with Williams' graduations in conjunction with an occlusal stent for the standardization of readings.

SECONDARY OUTCOMES:
Detect biochemically the nuclear factor kappa B (NF-κB) level in the gingival crevicular fluid (GCF). | Change from baseline to 1 month, from 1 month to 3 months, and from baseline to 3 months
  Levels of NF-κB (ng/ml) in GCF samples were determined by using a commercially available means of Enzyme Linked Immuno Sorbent Assay (ELISA) according to the manufacturer's recommendations. The GCF samples were collected using perio-paper strips (Oraflow Inc., Smithtown, New York, USA). Perio-paper strips visually contaminated with blood were discarded. The samples were immediately placed into a sterile, labeled Eppendorf tube and stored at -20 ºC for subsequent assays. Each perio-paper was soaked with 200ul of phosphate buffering saline (PBS), vortexed, and centrifuged. A supernatant was used for the detection of NF-κB. The kit was provided by Bioassay Technology Laboratory (China) Cat No E7121 Hu.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abuelela, Professor, Study Director — Professor of Oral medicine, Periodontology, and Oral Diagnosis, Faculty of Dentistry, Ain Shams University, Egypt; Olfat Shaker, Professor, Study Director — Professor of Medical Biochemistry and Molecular Biology, Faculty of Medicine, Cairo university, Egypt; Dina Osman, Professor, Study Director — Professor of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy (Girls), Al Azhar university, Egypt; Suzan Sarhan, PHD, Study Director — Lecturer of Oral Medicine, Periodontology, and Oral Diagnosis, Faculty of Dentistry, Ain Shams University, Egypt
Locations (1):
- Faculty of Dentitry, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Abouleish AE, Leib ML, Cohen NH. ASA provides examples to each ASA physical status class. ASA Monitor. 2015 Jun;79(6):38-49.
- [Background] Agarwal S, Chaubey KK, Chaubey A, Agarwal V, Madan E, Agarwal MC. Clinical efficacy of subgingivally delivered simvastatin gel in chronic periodontitis patients. J Indian Soc Periodontol. 2016 Jul-Aug;20(4):409-416. doi: 10.4103/0972-124X.194270. PMID 28298823
- [Background] Arunachalam R, Rajeev V, Vedam V, Ganapathy S, Dhanavel J . -Perioceutics in the management of Periodontal Disease.‖ J Young Pharm.;9(1):8-13., 2017
- [Background] Bansal M, Mittal N, Yadav SK, Khan G, Gupta P, Mishra B, Nath G. Periodontal thermoresponsive, mucoadhesive dual antimicrobial loaded in-situ gel for the treatment of periodontal disease: Preparation, in-vitro characterization and antimicrobial study. J Oral Biol Craniofac Res. 2018 May-Aug;8(2):126-133. doi: 10.1016/j.jobcr.2017.12.005. Epub 2017 Dec 13. PMID 29892535
- [Background] Juma Ab. The effects of Lepidium sativum seeds on fracture-induced healing in rabbits. MedGenMed. 2007 Apr 30;9(2):23. PMID 17955079
- [Background] Birkedal-Hansen H. Role of matrix metalloproteinases in human periodontal diseases. J Periodontol. 1993 May;64(5 Suppl):474-84. doi: 10.1902/jop.1993.64.5s.474. PMID 8315570
- [Background] Bostanci N, Ilgenli T, Emingil G, Afacan B, Han B, Toz H, Atilla G, Hughes FJ, Belibasakis GN. Gingival crevicular fluid levels of RANKL and OPG in periodontal diseases: implications of their relative ratio. J Clin Periodontol. 2007 May;34(5):370-6. doi: 10.1111/j.1600-051X.2007.01061.x. Epub 2007 Mar 13. PMID 17355365
- [Background] Aberg CH, Kelk P, Johansson A. Aggregatibacter actinomycetemcomitans: virulence of its leukotoxin and association with aggressive periodontitis. Virulence. 2015;6(3):188-95. doi: 10.4161/21505594.2014.982428. PMID 25494963
- [Background] Chakraborty A, Bhattacharjee A, Dasgupta P, Manna D, Chun WO. Simple Method for Standardization and Quantification of Linoleic Acid in Solanumnigrum Berries by HPTLC. Journal of Chromatography Separation Techniques. 2016;7:6.
- [Background] Donos N, Calciolari E, Brusselaers N, Goldoni M, Bostanci N, Belibasakis GN. The adjunctive use of host modulators in non-surgical periodontal therapy. A systematic review of randomized, placebo-controlled clinical studies. J Clin Periodontol. 2020 Jul;47 Suppl 22:199-238. doi: 10.1111/jcpe.13232. PMID 31834951
- [Background] El Kilani NS, Hazzaa HH, Hemoud HES, Imam O. Clinical and Radiographic Assessment of Single or Combined Treatment with Lepidium sativum and Alendronate of Non-Surgically Treated Chronic Periodontitis in Postmenopausal Osteoporotic Women. J Int Acad Periodontol. 2019 Jan 31;21(1):20-28. PMID 31522159
- [Background] Elhennawy E, Hammad A, Bilal M. Effect of Adjunctive Use of Simvastatin Gel in Management of Periodontitis on the Crevicular Fluid Calproteins Levels. Egyptian Dental Journal. 2022 Apr 1;68(2):1455-64.
- [Background] Euzebio Alves VT, de Andrade AK, Toaliar JM, Conde MC, Zezell DM, Cai S, Pannuti CM, De Micheli G. Clinical and microbiological evaluation of high intensity diode laser adjutant to non-surgical periodontal treatment: a 6-month clinical trial. Clin Oral Investig. 2013 Jan;17(1):87-95. doi: 10.1007/s00784-012-0703-7. Epub 2012 Mar 9. PMID 22402617
- [Background] Garala K, Joshi P, Shah M, Ramkishan A, Patel J. Formulation and evaluation of periodontal in situ gel. Int J Pharm Investig. 2013 Jan;3(1):29-41. doi: 10.4103/2230-973X.108961. PMID 23799203
- [Background] Gheorghe DN, Popescu DM, Salan A, Boldeanu MV, Ionele CM, Pitru A, Turcu-Stiolica A, Camen A, Florescu C, Rogoveanu I, Surlin P. Non-Surgical Periodontal Therapy Could Improve the Periodontal Inflammatory Status in Patients with Periodontitis and Chronic Hepatitis C. J Clin Med. 2021 Nov 13;10(22):5275. doi: 10.3390/jcm10225275. PMID 34830557
- [Background] Hajishengallis G, Wang M, Liang S. Induction of distinct TLR2-mediated proinflammatory and proadhesive signaling pathways in response to Porphyromonas gingivalis fimbriae. J Immunol. 2009 Jun 1;182(11):6690-6. doi: 10.4049/jimmunol.0900524. PMID 19454663
- [Background] Khurshid Z, Mali M, Naseem M, Najeeb S, Zafar MS. Human Gingival Crevicular Fluids (GCF) Proteomics: An Overview. Dent J (Basel). 2017 Feb 22;5(1):12. doi: 10.3390/dj5010012. PMID 29563418
- [Background] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. 2018 Jun;45 Suppl 20:S149-S161. doi: 10.1111/jcpe.12945. PMID 29926495
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Cobb CM. Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing. J Clin Periodontol. 2002 May;29 Suppl 2:6-16. PMID 12010523
- [Background] Pragati S, Ashok S, Kuldeep S. Recent advances in periodontal drug delivery systems. International Journal of Drug Delivery. 2009;1:1-9.
- [Background] Cicek Ari V, Ilarslan YD, Erman B, Sarkarati B, Tezcan I, Karabulut E, Oz SG, Tanriover MD, Sengun D, Berker E. Statins and IL-1beta, IL-10, and MPO Levels in Gingival Crevicular Fluid: Preliminary Results. Inflammation. 2016 Aug;39(4):1547-57. doi: 10.1007/s10753-016-0390-7. PMID 27290718
- [Background] Estanislau IM, Terceiro IR, Lisboa MR, Teles Pde B, Carvalho Rde S, Martins RS, Moreira MM. Pleiotropic effects of statins on the treatment of chronic periodontitis--a systematic review. Br J Clin Pharmacol. 2015 Jun;79(6):877-85. doi: 10.1111/bcp.12564. PMID 25444240
- [Background] Zeiser R. Immune modulatory effects of statins. Immunology. 2018 May;154(1):69-75. doi: 10.1111/imm.12902. Epub 2018 Feb 20. PMID 29392731
- [Background] Moro MG, Silveira Souto ML, Franco GCN, Holzhausen M, Pannuti CM. Efficacy of local phytotherapy in the nonsurgical treatment of periodontal disease: A systematic review. J Periodontal Res. 2018 Jun;53(3):288-297. doi: 10.1111/jre.12525. Epub 2018 Jan 19. PMID 29352465
- [Background] Rahman MA, Mossa JS, Al-Said MS, Al-Yahya MA. Medicinal plant diversity in the flora of Saudi Arabia 1: a report on seven plant families. Fitoterapia. 2004 Mar;75(2):149-61. doi: 10.1016/j.fitote.2003.12.012. PMID 15030919
- [Background] Pahla M, Moyo S, Muzemu T. Evaluating the effectiveness of botanical sprays in controlling Aphids (Brevicoryne brassicae) on rape (Brassica napus L.). International Journal of Agronomy and Agricultural Research. 2014;5(1):1-6.
- [Background] Prajapati VD, Maheriya PM, Jani GK, Patil PD, Patel BN. Lepidium sativum Linn.: a current addition to the family of mucilage and its applications. Int J Biol Macromol. 2014 Apr;65:72-80. doi: 10.1016/j.ijbiomac.2014.01.008. Epub 2014 Jan 10. PMID 24418343
- [Background] Sharma S, Agarwal N. Nourishing and healing prowess of garden cress (Lepidium sativum Linn.)-A review. 2011.
- [Background] Doke SGM. Garden cress (Lepidium sativum L.) seed-an important medicinal source: a review. J Nat Prod Plant Resour. 2014;4:69-80.
- [Background] Al-Sheddi ES, Farshori NN, Al-Oqail MM, Musarrat J, Al-Khedhairy AA, Siddiqui MA. Protective effect of Lepidium sativum seed extract against hydrogen peroxide-induced cytotoxicity and oxidative stress in human liver cells (HepG2). Pharm Biol. 2016;54(2):314-21. doi: 10.3109/13880209.2015.1035795. Epub 2015 Apr 17. PMID 25885937
- [Background] Raish M, Ahmad A, Alkharfy KM, Ahamad SR, Mohsin K, Al-Jenoobi FI, Al-Mohizea AM, Ansari MA. Hepatoprotective activity of Lepidium sativum seeds against D-galactosamine/lipopolysaccharide induced hepatotoxicity in animal model. BMC Complement Altern Med. 2016 Dec 3;16(1):501. doi: 10.1186/s12906-016-1483-4. PMID 27912738
- [Background] Rahman I. The role of oxidative stress in the pathogenesis of COPD: implications for therapy. Treat Respir Med. 2005;4(3):175-200. doi: 10.2165/00151829-200504030-00003. PMID 15987234
- [Background] Yadav YC, Srivastav DN, Seth AK. In vivo antioxidant potential of Lepidium sativum L. seeds in albino rats using cisplatin induced nephrotoxicity. Interact J Phytomed. 2010;2:292-8.
- [Background] Lang NP, Bartold PM. Periodontal health. J Periodontol. 2018 Jun;89 Suppl 1:S9-S16. doi: 10.1002/JPER.16-0517. PMID 29926938
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Fine DH, Patil AG, Loos BG. Classification and diagnosis of aggressive periodontitis. J Clin Periodontol. 2018 Jun;45 Suppl 20:S95-S111. doi: 10.1111/jcpe.12942. PMID 29926487
- [Background] Billings M, Holtfreter B, Papapanou PN, Mitnik GL, Kocher T, Dye BA. Age-dependent distribution of periodontitis in two countries: Findings from NHANES 2009 to 2014 and SHIP-TREND 2008 to 2012. J Clin Periodontol. 2018 Jun;45 Suppl 20:S130-S148. doi: 10.1111/jcpe.12944. PMID 29926501
- [Background] Needleman I, Garcia R, Gkranias N, Kirkwood KL, Kocher T, Iorio AD, Moreno F, Petrie A. Mean annual attachment, bone level, and tooth loss: A systematic review. J Clin Periodontol. 2018 Jun;45 Suppl 20:S112-S129. doi: 10.1111/jcpe.12943. PMID 29926483
- [Background] Hajishengallis G, Lamont RJ. Breaking bad: manipulation of the host response by Porphyromonas gingivalis. Eur J Immunol. 2014 Feb;44(2):328-38. doi: 10.1002/eji.201344202. PMID 24338806
- [Background] Sanz M, Beighton D, Curtis MA, Cury JA, Dige I, Dommisch H, Ellwood R, Giacaman RA, Herrera D, Herzberg MC, Kononen E, Marsh PD, Meyle J, Mira A, Molina A, Mombelli A, Quirynen M, Reynolds EC, Shapira L, Zaura E. Role of microbial biofilms in the maintenance of oral health and in the development of dental caries and periodontal diseases. Consensus report of group 1 of the Joint EFP/ORCA workshop on the boundaries between caries and periodontal disease. J Clin Periodontol. 2017 Mar;44 Suppl 18:S5-S11. doi: 10.1111/jcpe.12682. PMID 28266109
- [Background] Preshaw PM, Taylor JJ. How has research into cytokine interactions and their role in driving immune responses impacted our understanding of periodontitis? J Clin Periodontol. 2011 Mar;38 Suppl 11:60-84. doi: 10.1111/j.1600-051X.2010.01671.x. PMID 21323705
- [Background] Cekici A, Kantarci A, Hasturk H, Van Dyke TE. Inflammatory and immune pathways in the pathogenesis of periodontal disease. Periodontol 2000. 2014 Feb;64(1):57-80. doi: 10.1111/prd.12002. PMID 24320956
- [Background] Kinane DF, Preshaw PM, Loos BG; Working Group 2 of Seventh European Workshop on Periodontology. Host-response: understanding the cellular and molecular mechanisms of host-microbial interactions--consensus of the Seventh European Workshop on Periodontology. J Clin Periodontol. 2011 Mar;38 Suppl 11:44-8. doi: 10.1111/j.1600-051X.2010.01682.x. PMID 21323703
- [Background] Olsen I, Lambris JD, Hajishengallis G. Porphyromonas gingivalis disturbs host-commensal homeostasis by changing complement function. J Oral Microbiol. 2017 Jun 30;9(1):1340085. doi: 10.1080/20002297.2017.1340085. eCollection 2017. PMID 28748042
- [Background] Crotti T, Smith MD, Hirsch R, Soukoulis S, Weedon H, Capone M, Ahern MJ, Haynes D. Receptor activator NF kappaB ligand (RANKL) and osteoprotegerin (OPG) protein expression in periodontitis. J Periodontal Res. 2003 Aug;38(4):380-7. doi: 10.1034/j.1600-0765.2003.00615.x. PMID 12828654
- [Background] Chapple IL, Brock GR, Milward MR, Ling N, Matthews JB. Compromised GCF total antioxidant capacity in periodontitis: cause or effect? J Clin Periodontol. 2007 Feb;34(2):103-10. doi: 10.1111/j.1600-051X.2006.01029.x. Epub 2006 Dec 13. PMID 17214737
- [Background] Golz L, Memmert S, Rath-Deschner B, Jager A, Appel T, Baumgarten G, Gotz W, Frede S. Hypoxia and P. gingivalis synergistically induce HIF-1 and NF-kappaB activation in PDL cells and periodontal diseases. Mediators Inflamm. 2015;2015:438085. doi: 10.1155/2015/438085. Epub 2015 Mar 15. PMID 25861162
- [Background] Ambili R, Janam P. A critique on nuclear factor-kappa B and signal transducer and activator of transcription 3: The key transcription factors in periodontal pathogenesis. J Indian Soc Periodontol. 2017 Sep-Oct;21(5):350-356. doi: 10.4103/jisp.jisp_301_16. PMID 29491579
- [Background] Chang J, Wang Z, Tang E, Fan Z, McCauley L, Franceschi R, Guan K, Krebsbach PH, Wang CY. Inhibition of osteoblastic bone formation by nuclear factor-kappaB. Nat Med. 2009 Jun;15(6):682-9. doi: 10.1038/nm.1954. PMID 19448637
- [Background] Chen X, Hu C, Wang G, Li L, Kong X, Ding Y, Jin Y. Nuclear factor-kappaB modulates osteogenesis of periodontal ligament stem cells through competition with beta-catenin signaling in inflammatory microenvironments. Cell Death Dis. 2013 Feb 28;4(2):e510. doi: 10.1038/cddis.2013.14. PMID 23449446
- [Background] Smiley CJ, Tracy SL, Abt E, Michalowicz BS, John MT, Gunsolley J, Cobb CM, Rossmann J, Harrel SK, Forrest JL, Hujoel PP, Noraian KW, Greenwell H, Frantsve-Hawley J, Estrich C, Hanson N. Systematic review and meta-analysis on the nonsurgical treatment of chronic periodontitis by means of scaling and root planing with or without adjuncts. J Am Dent Assoc. 2015 Jul;146(7):508-24.e5. doi: 10.1016/j.adaj.2015.01.028. PMID 26113099
- [Background] Graziani F, Karapetsa D, Alonso B, Herrera D. Nonsurgical and surgical treatment of periodontitis: how many options for one disease? Periodontol 2000. 2017 Oct;75(1):152-188. doi: 10.1111/prd.12201. PMID 28758300
- [Background] Ehizele A, Akhionbare O. Effect of non-surgical periodontal therapy on the concentration of volatile sulfur compound in mouth air of a group of nigerian young adults. Ann Med Health Sci Res. 2013 Jul;3(3):433-7. doi: 10.4103/2141-9248.117951. PMID 24116328
- [Background] Keestra JA, Grosjean I, Coucke W, Quirynen M, Teughels W. Non-surgical periodontal therapy with systemic antibiotics in patients with untreated chronic periodontitis: a systematic review and meta-analysis. J Periodontal Res. 2015 Jun;50(3):294-314. doi: 10.1111/jre.12221. Epub 2014 Aug 21. PMID 25142259
- [Background] Zandbergen D, Slot DE, Niederman R, Van der Weijden FA. The concomitant administration of systemic amoxicillin and metronidazole compared to scaling and root planing alone in treating periodontitis: =a systematic review=. BMC Oral Health. 2016 Feb 29;16:27. doi: 10.1186/s12903-015-0123-6. PMID 26928597
- [Background] Caton JG, Ciancio SG, Blieden TM, Bradshaw M, Crout RJ, Hefti AF, Massaro JM, Polson AM, Thomas J, Walker C. Treatment with subantimicrobial dose doxycycline improves the efficacy of scaling and root planing in patients with adult periodontitis. J Periodontol. 2000 Apr;71(4):521-32. doi: 10.1902/jop.2000.71.4.521. PMID 10807113
- [Background] Herrera D, Matesanz P, Bascones-Martinez A, Sanz M. Local and systemic antimicrobial therapy in periodontics. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):50-60. doi: 10.1016/S1532-3382(12)70013-1. PMID 23040339
- [Background] Preshaw PM, Novak MJ, Mellonig J, Magnusson I, Polson A, Giannobile WV, Rowland RW, Thomas J, Walker C, Dawson DR, Sharkey D, Bradshaw MH. Modified-release subantimicrobial dose doxycycline enhances scaling and root planing in subjects with periodontal disease. J Periodontol. 2008 Mar;79(3):440-52. doi: 10.1902/jop.2008.070375. PMID 18315426
- [Background] H R R, Dhamecha D, Jagwani S, Rao M, Jadhav K, Shaikh S, Puzhankara L, Jalalpure S. Local drug delivery systems in the management of periodontitis: A scientific review. J Control Release. 2019 Aug 10;307:393-409. doi: 10.1016/j.jconrel.2019.06.038. Epub 2019 Jun 27. PMID 31255689
- [Background] Kaplish V, Walia MK, Kumar HS. Local drug delivery systems in the treatment of periodontitis:A review. Pharmacophore. 2013;4:39-49.
- [Background] Han JY, Reynolds MA. Effect of anti-rheumatic agents on periodontal parameters and biomarkers of inflammation: a systematic review and meta-analysis. J Periodontal Implant Sci. 2012 Feb;42(1):3-12. doi: 10.5051/jpis.2012.42.1.3. Epub 2012 Feb 29. PMID 22413068
- [Background] Lamster IB. Evaluation of components of gingival crevicular fluid as diagnostic tests. Ann Periodontol. 1997 Mar;2(1):123-37. doi: 10.1902/annals.1997.2.1.123. PMID 9151549
- [Background] Sachdeva S, Agarwal V. Evaluation of commercially available biodegradable tetracycline fiber therapy in chronic periodontitis. J Indian Soc Periodontol. 2011 Apr;15(2):130-4. doi: 10.4103/0972-124X.84381. PMID 21976836
- [Background] Chhina S, Rathore AS, Juneja S. Alpha-2-Macroglobulin Levels in Gingival Crevicular Fluid Pre- and Post-scaling and Root Planing with Adjunctive Tetracycline Fibers in Chronic Periodontitis: A Randomized Controlled Trial. J Contemp Dent Pract. 2015 Jun 1;16(6):474-8. doi: 10.5005/jp-journals-10024-1709. PMID 26323451
- [Background] Khan FY, Jan SM, Mushtaq M. Clinical utility of locally-delivered collagen-based biodegradable tetracycline fibers in periodontal therapy: an in vivo study. J Investig Clin Dent. 2015 Nov;6(4):307-12. doi: 10.1111/jicd.12111. Epub 2014 Jul 17. PMID 25044345
- [Result] 1.Abdelghany AM, El-Damrawi G, Oraby AH, Madshal MA. Optical and FTIR structural studies on CoO-doped strontium phosphate glasses. Journal of Non-Crystalline Solids. 2018 Nov 1;499:153-8.
- [Result] 2.Abdel-Hameed HS, El-Saeed SM, Ahmed NS, Nassar AM, El-Kafrawy AF, Hashem AI. Chemical transformation of Jojoba oil and Soybean oil and study of their uses as bio-lubricants. Industrial Crops and Products. 2022 Nov 1;187:115256.